CLINICAL TRIAL: NCT02454231
Title: Monocentric Randomized Study for the Therapy of Critic Limb Ischemia With Bone Marrow- or Peripheral Blood-derived Stem Cells
Brief Title: Monocentric Trial: Stem Cell Emergency Life Threatening Limbs Arteriopathy (SCELTA)
Acronym: SCELTA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florence (Other)
Collaborators: Tuscany Region (Unknown)
Responsible Party: Principal Investigator, Enrico Maggi, Professor, MD, Director of the Unit of Immunology and Cellular Therapy, University of Florence
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFlorence
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Critical Limb Ischemia
Keywords: EPC; CD34+; CD14+CD34low
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peripheral blood EPC injection (Experimental)
  Interventions: Biological: Transplantation of circulating CD14+CD34+cells
- bone marrow MNC injection (Active Comparator)
  Interventions: Biological: Transplantation of BM MNC

INTERVENTIONS:
Biological: Transplantation of circulating CD14+CD34+cells — intramuscular injection of circulating EPC at leg level
  Arms: peripheral blood EPC injection
Biological: Transplantation of BM MNC — intramuscular injection of BM MNC at leg level
  Arms: bone marrow MNC injection

SUMMARY:
The investigators designed a randomized clinical trial (stem cell emergency life threatening arteriopathy or SCELTA) to compare the therapeutic efficacy of the auto-transplant of enriched circulating EPCs (ECEPCs) with auto-transplant of BM-MNCs. ECEPCs, obtained by immunoselection of CD14+ and CD34+ cells, or BM-MNCs, were injected intramuscularly in the affected limb of patients with critical limb ischemia (CLI).

DETAILED DESCRIPTION:
Peripheral arterial disease comprises a clinical spectrum that extends from no symptoms to presentation with critical limb ischemia (CLI), which is a very invalidating condition characterized by rest pain, march inability, trophic lesions and unavoidable progression to major amputations, which are burdened by a high mortality in the first year. The pathophysiology of CLI often associates with a defect in the development of collateral vessels and angiogenesis, a process which refers to the formation of new blood vessels into tissue, due to circulating endothelial progenitor cells (EPCs) and vascular progenitor cells. In the last few years, significant improvement of this condition has been reported following bone marrow (BM) autotransplant or autotransplant of peripheral EPCs mobilized from BM through the injection of granulocyte-colony stimulatory factor (G-CSF). In a previous study, the investigators found that individually variable proportions of circulating CD14+ cells expressed low levels of CD34 (CD14+CD34low) and revealed the functional phenotype of EPCs. The investigators therefore designed a monocentric randomized clinical trial to compare the therapeutic efficacy of BM autotransplant with the autotransplant of a population of circulating CD34+ and CD14+CD34low enriched by a closed sterile immunomagnetic system (enriched circulating EPCs or ECEPCs), without a previous EPC mobilization from BM.

Patients will be evaluated for clinical parameters and ABI, TBI, TCp02 before autotransplant and at three follow-up times after the autotransplant (4, 24 and 52 weeks); also angio-TAC of legs, capillaroscopy, and photoplethysmography will be evaluated at 4, and even at 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were men and women aged more than 40 years with a diagnosis of CLI due to atherosclerosis of the lower extremities, as defined by the presence of persistent rest pain requiring systemic and continued analgesic treatment in the last 15 days and/or the presence of trophic lesions imputable to the occluding arteriopathy, an ankle-brachial Index (ABI) < 0.40 (with systolic ankle pressure < 50-70 Hg mm), a toe/brachial index (TBI) < 0.40 (with big toe systolic pressure < 30-50 Hg mm), and a transcutaneous oxygen pressure (TC pO2) < 30 Hg mm.
* The patient was considered as eligible for the treatment and enrolled only after the demonstration that intravascular or surgical re-vascularization was not possible, as revealed by ecography and angio-CAT, or when the patient refused to undergo surgical treatments and after having obtained his/her written informed consensus.

Exclusion Criteria:

* Exclusion criteria were: age < 40;
* not atherosclerotic CLI,
* myocardial infarction occurrence in the 6 months;
* cardiac failure of III-IV class NYHA;
* ejection fraction lower than 40%;
* arterial hypertension (>160/100 Hg mm) uncontrolled despite the usage of two anti-hypertensive drugs;
* presence of current or chronic severe infectious diseases;
* osteomyelitis;
* diabetes with glycate hemoglobin > 7.5;
* proliferative diabetic retinopathy;
* hemorrhagic disorders;
* non-atherosclerotic arteriopathy;
* chronic airway insufficiency (p02 <65 Hg mm, pCO2 > 0.50 Hg mm);
* renal failure (creatinine > 2mg/dl);
* contraindications or intolerance to contrast media for radiologic imaging

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-09; Primary Completion 2015-05 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety as measured by evaluation of any adverse event temporary correlated with the treatment | 52 weeks of follow-up
  Evaluation of any adverse event temporary correlated with the treatment
Changes in ischemic leg perfusion from baseline | 4, 22, 52 weeks of follow-up
  Improvement of leg perfusion as assessed by values of Time to Pick (TTP) evaluated by ultrasound tools

SECONDARY OUTCOMES:
Improvement of Mean values of the transcutaneous partial oxygen pressure (TCP02) | 4, 22, 52 weeks of follow-up
  Improvement of mean values of the transcutaneous partial oxygen pressure of at least 20%
Improvement of mean values of ankle brachial pressure index (ABI) | 4, 22, 52 weeks of follow-up
  improvement (at least 25% increase) of Mean values of ankle brachial pressure index
Improvement of vessel anatomical status | 4, 22, 52 weeks of follow-up
  Improvement of leg vascularization as assessed by color Doppler ultrasound
Improvement of leg perfusion | 4, 22, 52 weeks of follow-up
  Improvement of leg perfusion as assessed by plethysmography characterization
Improvement of vessel anatomical status | 4, 22, 52 weeks of follow-up
  Improvement of leg vascularization as assessed by Angio-CT, defined as presence of new vessels
Quality of life Improvement | -28, 0, 28 weeks of follow-up
  Quality of life, as assessed by the disease-specific ST22 and SF36 questionaries
improvement of rest pain | 4, 22, 52 weeks of follow-up
  Rest pain as evaluated by visual analogue pain scale (VAS)
Improvement of trophic limb lesions | 4, 22, 52 weeks of follow-up
  Mean score of trophic limb lesions, as evaluated according to Wagner international grade
Reduction of numbers of major amputation (amputation free survival ) | 4, 22, 52 weeks of follow-up
  Reduction of numbers of major amputation compared with untreated patients
improvement of microvascular anatomy | 4, 22, 52 weeks of follow-up
  evaluation of microvascular anatomy as assessed by capillaroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Maggi, professor, Principal Investigator — University of Florence
Locations (1):
- Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany, Italy

REFERENCES:
- [Background] Weitz JI, Byrne J, Clagett GP, Farkouh ME, Porter JM, Sackett DL, Strandness DE Jr, Taylor LM. Diagnosis and treatment of chronic arterial insufficiency of the lower extremities: a critical review. Circulation. 1996 Dec 1;94(11):3026-49. doi: 10.1161/01.cir.94.11.3026. No abstract available. PMID 8941154
- [Background] Gregg EW, Sorlie P, Paulose-Ram R, Gu Q, Eberhardt MS, Wolz M, Burt V, Curtin L, Engelgau M, Geiss L; 1999-2000 national health and nutrition examination survey. Prevalence of lower-extremity disease in the US adult population >=40 years of age with and without diabetes: 1999-2000 national health and nutrition examination survey. Diabetes Care. 2004 Jul;27(7):1591-7. doi: 10.2337/diacare.27.7.1591. PMID 15220233
- [Background] Curb JD, Masaki K, Rodriguez BL, Abbott RD, Burchfiel CM, Chen R, Petrovitch H, Sharp D, Yano K. Peripheral artery disease and cardiovascular risk factors in the elderly. The Honolulu Heart Program. Arterioscler Thromb Vasc Biol. 1996 Dec;16(12):1495-500. doi: 10.1161/01.atv.16.12.1495. PMID 8977454
- [Background] Meijer WT, Grobbee DE, Hunink MG, Hofman A, Hoes AW. Determinants of peripheral arterial disease in the elderly: the Rotterdam study. Arch Intern Med. 2000 Oct 23;160(19):2934-8. doi: 10.1001/archinte.160.19.2934. PMID 11041900
- [Background] Melillo E, Nuti M, Bongiorni L, Golgini E, Balbarini A. [Major and minor amputation rates and lower critical limb ischemia: the epidemiological data of western Tuscany]. Ital Heart J Suppl. 2004 Oct;5(10):794-805. Italian. PMID 15615351
- [Background] Inglese L, Graziani L, Tarricone R. [Percutaneous treatment of peripheral obstructive arteriopathy: the reasons for a choice]. Ital Heart J Suppl. 2000 Sep;1(9):1138-47. Italian. PMID 11140282
- [Background] Dzau VJ, Gnecchi M, Pachori AS, Morello F, Melo LG. Therapeutic potential of endothelial progenitor cells in cardiovascular diseases. Hypertension. 2005 Jul;46(1):7-18. doi: 10.1161/01.HYP.0000168923.92885.f7. Epub 2005 Jun 13. PMID 15956118
- [Background] Ikenaga S, Hamano K, Nishida M, Kobayashi T, Li TS, Kobayashi S, Matsuzaki M, Zempo N, Esato K. Autologous bone marrow implantation induced angiogenesis and improved deteriorated exercise capacity in a rat ischemic hindlimb model. J Surg Res. 2001 Apr;96(2):277-83. doi: 10.1006/jsre.2000.6080. PMID 11266284
- [Background] Kalka C, Masuda H, Takahashi T, Kalka-Moll WM, Silver M, Kearney M, Li T, Isner JM, Asahara T. Transplantation of ex vivo expanded endothelial progenitor cells for therapeutic neovascularization. Proc Natl Acad Sci U S A. 2000 Mar 28;97(7):3422-7. doi: 10.1073/pnas.97.7.3422. PMID 10725398
- [Background] Iwaguro H, Yamaguchi J, Kalka C, Murasawa S, Masuda H, Hayashi S, Silver M, Li T, Isner JM, Asahara T. Endothelial progenitor cell vascular endothelial growth factor gene transfer for vascular regeneration. Circulation. 2002 Feb 12;105(6):732-8. doi: 10.1161/hc0602.103673. PMID 11839630
- [Background] Iba O, Matsubara H, Nozawa Y, Fujiyama S, Amano K, Mori Y, Kojima H, Iwasaka T. Angiogenesis by implantation of peripheral blood mononuclear cells and platelets into ischemic limbs. Circulation. 2002 Oct 8;106(15):2019-25. doi: 10.1161/01.cir.0000031332.45480.79. PMID 12370229 (Retraction: PMID 23704253 Circulation. 2013 Jun 11;127(23):e842)
- [Background] Tateishi-Yuyama E, Matsubara H, Murohara T, Ikeda U, Shintani S, Masaki H, Amano K, Kishimoto Y, Yoshimoto K, Akashi H, Shimada K, Iwasaka T, Imaizumi T; Therapeutic Angiogenesis using Cell Transplantation (TACT) Study Investigators. Therapeutic angiogenesis for patients with limb ischaemia by autologous transplantation of bone-marrow cells: a pilot study and a randomised controlled trial. Lancet. 2002 Aug 10;360(9331):427-35. doi: 10.1016/S0140-6736(02)09670-8. PMID 12241713
- [Background] Masuda H, Asahara T. Post-natal endothelial progenitor cells for neovascularization in tissue regeneration. Cardiovasc Res. 2003 May 1;58(2):390-8. doi: 10.1016/s0008-6363(02)00785-x. PMID 12757873
- [Background] Romagnani P, Annunziato F, Liotta F, Lazzeri E, Mazzinghi B, Frosali F, Cosmi L, Maggi L, Lasagni L, Scheffold A, Kruger M, Dimmeler S, Marra F, Gensini G, Maggi E, Romagnani S. CD14+CD34low cells with stem cell phenotypic and functional features are the major source of circulating endothelial progenitors. Circ Res. 2005 Aug 19;97(4):314-22. doi: 10.1161/01.RES.0000177670.72216.9b. Epub 2005 Jul 14. PMID 16020753
- [Background] Chambers I, Colby D, Robertson M, Nichols J, Lee S, Tweedie S, Smith A. Functional expression cloning of Nanog, a pluripotency sustaining factor in embryonic stem cells. Cell. 2003 May 30;113(5):643-55. doi: 10.1016/s0092-8674(03)00392-1. PMID 12787505
- [Background] Mitsui K, Tokuzawa Y, Itoh H, Segawa K, Murakami M, Takahashi K, Maruyama M, Maeda M, Yamanaka S. The homeoprotein Nanog is required for maintenance of pluripotency in mouse epiblast and ES cells. Cell. 2003 May 30;113(5):631-42. doi: 10.1016/s0092-8674(03)00393-3. PMID 12787504
- [Background] Pesce M, Scholer HR. Oct-4: gatekeeper in the beginnings of mammalian development. Stem Cells. 2001;19(4):271-8. doi: 10.1634/stemcells.19-4-271. PMID 11463946
- [Background] Iwama A, Oguro H, Negishi M, Kato Y, Morita Y, Tsukui H, Ema H, Kamijo T, Katoh-Fukui Y, Koseki H, van Lohuizen M, Nakauchi H. Enhanced self-renewal of hematopoietic stem cells mediated by the polycomb gene product Bmi-1. Immunity. 2004 Dec;21(6):843-51. doi: 10.1016/j.immuni.2004.11.004. PMID 15589172
- [Background] Melillo E, Ferrari M, Balbarini A, Pedrinelli R. Transcutaneous gases determination in diabetic critical limb ischemia. Diabetes Care. 2005 Aug;28(8):2081-2. doi: 10.2337/diacare.28.8.2081. No abstract available. PMID 16043766
- [Background] Becker F, Gabrielle F, Raoux MH, Brenot R, David M. [Value of measuring transcutaneous oxygen pressure in arterial disease of the legs]. Ann Cardiol Angeiol (Paris). 1989 Oct;38(8):465-72. French. PMID 2596817